CLINICAL TRIAL: NCT00003378
Title: A Phase I Feasibility Trial of Carboplatin, Paclitaxel, and Gemcitabine in Patients With Previously Untreated Epithelial Ovarian Carcinoma and Primary Peritoneal Carcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Previously Untreated Stage III or Stage IV Ovarian or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000066372; GOG-9801
Record Dates: First submitted 1999-11-01; First posted 2004-08-26 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2011-12

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Gemcitabine; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy in treating patients with previously untreated stage III or stage IV ovarian or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of administering multiple courses of chemotherapy without excessive dose modification or treatment delay in patients with previously untreated ovarian epithelial carcinoma or primary peritoneal carcinoma. II. Determine the response rate (in patients with measurable disease) and progression-free interval in these patients receiving this treatment.

OUTLINE: This is a feasibility study. On day 1, patients receive paclitaxel as a 3 hour continuous IV infusion followed by carboplatin as a 30 minute infusion. Gemcitabine is administered by continuous infusion over 30 minutes on day 1 following carboplatin and on day 8. In the absence of disease progression or unacceptable toxicity, courses repeat every 21 days for a maximum of 8 courses. Patients are followed every 3 months for 2 years, every 6 months for the next 3 years, and annually thereafter.

PROJECTED ACCRUAL: A total of 15-45 patients will be accrued for this study within approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, previously untreated: Stage III or stage IV ovarian epithelial cancer Stage III or stage IV primary peritoneal cancer

PATIENT CHARACTERISTICS: Age: 18 to 80 Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 3 times ULN Alkaline phosphatase no greater than 3 times ULN Renal: Creatinine no greater than 1.5 mg/dL Other: Effective contraception required of fertile patients No significant infections No other severe medical problems that would subject patient to undue risk from this protocol No other active malignancy within past 5 years except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for this or any other malignancy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for this or any other malignancy Surgery: No prior surgery other than cytoreductive surgery and recovered

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 1998-08; Primary Completion 2000-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Y. Look, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (64):
- United States (63):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Brookview Research, Inc., Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- NCIC-Clinical Trials Group, Kingston, Ontario, Canada

REFERENCES:
- [Result] Gould N, Sill MW, Mannel RS, Thaker PH, Disilvestro P, Waggoner S, Yamada SD, Armstrong DK, Wenzel L, Huang H, Fracasso PM, Walker JL. A phase I study with an expanded cohort to assess the feasibility of intravenous paclitaxel, intraperitoneal carboplatin and intraperitoneal paclitaxel in patients with untreated ovarian, fallopian tube or primary peritoneal carcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2012 Apr;125(1):54-8. doi: 10.1016/j.ygyno.2011.12.417. Epub 2011 Dec 11. PMID 22155262
- [Result] Look KY, Bookman MA, Schol J, Herzog TJ, Rocereto T, Vinters J; Gynecologic Oncology Group Study. Phase I feasibility trial of carboplatin, paclitaxel, and gemcitabine in patients with previously untreated epithelial ovarian or primary peritoneal cancer: a Gynecologic Oncology Group study. Gynecol Oncol. 2004 Jan;92(1):93-100. doi: 10.1016/j.ygyno.2003.09.019. PMID 14751144